CLINICAL TRIAL: NCT00725621
Title: Real Life Dosing Regimen of Remicade in Austria, Monitored Over 9 Consecutive Infusions in Rheumatoid Arthritis Therapy
Brief Title: Real Life Dosing of Remicade for Rheumatoid Arthritis in Austria Monitored Over 9 Infusions (Study P03756)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P03756
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remicade: Patients with severe RA (indication according to Austrian labeling) will receive Remicade induction therapy consisting of three Remicade infusions in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy will consist of another maximal 6 infusions. Remicade induction and maintenance therapy doses and intervals will be at the discretion of the physicians.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Remicade induction therapy consisting of three Remicade infusions in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy will consist of another maximal 6 infusions given in doses and intervals due to discretion of physicians.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is a prospective, open-label, 1-arm, multicenter observational study to determine the average Remicade dosage and time span between 9 infusions in subjects with rheumatoid arthritis (RA)

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* Severe RA (indication according to Austrian labeling).

Exclusion Criteria:

* According to Summary of Product Characteristics (SPC).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe RA being treated at specialized centers.
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2004-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Remicade (Specialized Hospitals & Extramural Infusion Centers): Remicade induction therapy consisted of 3 infusions (3 mg/kg) in weeks 0, 2, and 6 given in specialized centers (specialized hospitals and extramural infusion centers). Maintenance therapy consisted of a maximum of 6 infusions (3 mg/kg) given in doses and intervals at the discretion of physician. The observation period could not exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in Summary of Product Characteristics (SPC) was taken into consideration.
Period: Overall Study
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Started | 516 (Started was defined as the number of participants who received at least one infusion of Remicade.)
Completed | 245 (Completed was defined as the number of participants who received 9 consecutive Remicade infusions.)
Not Completed | 271
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 46
Not completed — Withdrawal by Subject | 57
Not completed — Physician Decision | 19
Not completed — Lost to Follow-up | 52
Not completed — Non-compliance | 8
Not completed — Continued treatment by other physician | 6
Not completed — Switched to other study | 1
Not completed — Switched to other drug | 1
Not completed — Prepared for elective surgery | 1
Not completed — Reason not specified | 55

BASELINE CHARACTERISTICS:
Groups:
- Remicade (Specialized Hospitals & Extramural Infusion Centers): Remicade induction therapy consisted of 3 infusions (3 mg/kg) in weeks 0, 2, and 6 given in specialized centers (specialized hospitals and extramural infusion centers). Maintenance therapy consisted of a maximum of 6 infusions (3 mg/kg) given in doses and intervals at the discretion of physician. The observation period could not exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in SPC was taken into consideration.
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Number analyzed (Participants) | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398
  Male | 118

OUTCOME MEASURES:

1. Primary Outcome: Mean Time Interval Between Remicade Infusions in Participants During Maintenance Treatment Following Induction Therapy
Description: The impact of the maintenance therapy location (specialized hospitals versus extramural infusion centers) was also examined.
Time Frame: Maximum of 16 weeks
Population: Remicade-naive participants who received Remicade induction therapy and subsequent maintenance therapy during the observational study.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Remicade (Specialized Hospitals Only): Remicade induction therapy consisted of 3 infusions (3 mg/kg) in weeks 0, 2, and 6 given in specialized hospitals. Maintenance therapy consisted of a maximum of 6 infusions (3 mg/kg) given in doses and intervals at the discretion of physician. The observation period could not exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in SPC was taken into consideration.
- Remicade (Extramural Infusion Centers Only): Remicade induction therapy consisted of 3 infusions (3 mg/kg) in weeks 0, 2, and 6 given in extramural infusion centers. Maintenance therapy consisted of a maximum of 6 infusions (3 mg/kg) given in doses and intervals at the discretion of physician. The observation period could not exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in SPC was taken into consideration.
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers) | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 193 | 120 | 73
Days
  Infusion 3/4 (n=193, n=120, n=73) | 56.48 (10.94) | 56.32 (7.76) | 56.75 (14.82)
  Infusion 4/5 (n=193, n=120, n=73) | 57.55 (10.81) | 56.83 (10.66) | 58.73 (11.03)
  Infusion 5/6 (n=178, n=110, n=68) | 56.80 (10.85) | 56.60 (13.07) | 57.13 (5.75)
  Infusion 6/7 (n=163, n=99, n=64) | 56.07 (8.57) | 55.41 (8.56) | 57.09 (8.56)
  Infusion 7/8 (n=153, n=91, n=62) | 57.33 (10.97) | 56.43 (12.11) | 58.65 (8.97)
  Infusion 8/9 (n=143, n=83, n=60) | 57.04 (11.07) | 56.60 (12.49) | 57.65 (8.80)

2. Primary Outcome: Median Time Interval Between Remicade Infusions in Participants During Maintenance Treatment Following Induction Therapy
Description: as for outcome 1
Time Frame: Maximum of 16 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers) | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 193 | 120 | 73
Days
  Infusion 3/4 (n=193, n=120, n=73) | 57.00 [25.00 to 135.00] | 57.00 [29.00 to 85.00] | 57.00 [25.00 to 135.00]
  Infusion 4/5 (n=193, n=120, n=73) | 57.00 [41.00 to 120.00] | 57.00 [41.00 to 116.00] | 57.00 [43.00 to 120.00]
  Infusion 5/6 (n=178, n=110, n=68) | 57.00 [30.00 to 140.00] | 57.00 [30.00 to 140.00] | 57.00 [42.00 to 71.00]
  Infusion 6/7 (n=163, n=99, n-64) | 57.00 [30.00 to 106.00] | 57.00 [41.00 to 92.00] | 57.00 [30.00 to 106.00]
  Infusion 7/8 (n=153, n=91, n=62) | 57.00 [13.00 to 112.00] | 57.00 [13.00 to 97.00] | 57.00 [44.00 to 112.00]
  Infusion 8/9 (n=143, n=83, n=60) | 57.00 [24.00 to 113.00] | 57.00 [24.00 to 113.00] | 57.00 [43.00 to 111.00]

3. Primary Outcome: Mean Dose of Remicade in Participants Receiving Induction Therapy and Subsequent Maintenance Therapy
Description: as for outcome 1
Time Frame: Maximum of 102 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/kilograms (mg/kg)
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers) | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 193 | 120 | 73
milligrams/kilograms (mg/kg)
  Infusion 1 (n=193, n=120, n=73) | 3.42 (0.59) | 3.50 (0.59) | 3.30 (0.56)
  Infusion 2 (n=192, n=119, n=73) | 3.43 (0.59) | 3.51 (0.59) | 3.31 (0.56)
  Infusion 3 (n=193, n=120, n=73) | 3.46 (0.62) | 3.56 (0.65) | 3.30 (0.54)
  Infusion 4 (n=193, n=120, n=73) | 3.50 (0.62) | 3.59 (0.63) | 3.36 (0.57)
  Infusion 5 (n=193, n=120, n=73) | 3.53 (0.67) | 3.62 (0.71) | 3.36 (0.58)
  Infusion 6 (n=178, n=110, n=68) | 3.56 (0.70) | 3.70 (0.75) | 3.34 (0.54)
  Infusion 7 (n=163, n=99, n=64) | 3.63 (0.74) | 3.78 (0.82) | 3.39 (0.53)
  Infusion 8 (n=153, n=91, n=62) | 3.60 (0.72) | 3.75 (0.79) | 3.37 (0.53)
  Infusion 9 (n=143, n=83, n=60) | 3.61 (0.72) | 3.79 (0.78) | 3.36 (0.54)

4. Secondary Outcome: Disease Progression Specified by the Time Period Between Onset of Rheumatoid Arthritis (RA) and Onset of Remicade Therapy
Time Frame: 24 months maximum
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Number analyzed (Participants) | 511
Years | 8.02 (8.07)

5. Secondary Outcome: Number and Kind of Previous Therapies With Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
Description: Some participants had more than one previous treatment with a DMARD.
Time Frame: 24 months maximum
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Number; unit: Participants
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Number analyzed (Participants) | 516
Participants
  Methotrexate | 470
  Sulfasalazine | 111
  Leflunomide | 138

6. Primary Outcome: Median Dose of Remicade in Participants Receiving Induction Therapy and Subsequent Maintenance Therapy
Description: as for outcome 1
Time Frame: Maximum of 102 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers) | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 193 | 120 | 73
mg/kg
  Infusion 1 (n=193, n=120, n=73) | 3.33 [2.25 to 6.15] | 3.38 [2.45 to 5.97] | 3.23 [2.25 to 6.15]
  Infusion 2 (n=192, n=119, n=73) | 3.33 [2.25 to 6.15] | 3.39 [2.56 to 5.97] | 3.23 [2.25 to 6.15]
  Infusion 3 (n=193, n=120, n=73) | 3.33 [2.22 to 5.97] | 3.40 [2.22 to 5.88] | 3.23 [2.41 to 5.97]
  Infusion 4 (n=193, n=120, n=73) | 3.41 [2.44 to 5.80] | 3.49 [2.50 to 5.80] | 3.33 [2.44 to 5.80]
  Infusion 5 (n=193, n=120, n=73) | 3.39 [2.08 to 5.71] | 3.53 [2.08 to 5.48] | 3.33 [2.35 to 5.71]
  Infusion 6 (n=178, n=110, n=68) | 3.41 [2.13 to 5.71] | 3.61 [2.13 to 5.48] | 3.33 [2.35 to 5.71]
  Infusion 7 (n=163, n=99, n=64) | 3.53 [2.13 to 5.71] | 3.70 [2.13 to 5.66] | 3.33 [2.56 to 5.71]
  Infusion 8 (n=153, n=91, n=62) | 3.53 [2.13 to 5.71] | 3.70 [2.13 to 5.56] | 3.33 [2.50 to 5.71]
  Infusion 9 (n=143, n=83, n=60) | 3.53 [2.38 to 5.71] | 3.70 [2.43 to 5.56] | 3.33 [2.38 to 5.71]

7. Primary Outcome: Mean Remicade Dose Per Participant
Time Frame: Maximum of 102 weeks
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Number analyzed (Participants) | 500
mg/kg | 3.56 (0.63)

8. Primary Outcome: Median Remicade Dose Per Participant
Time Frame: Maximum of 102 weeks
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Number analyzed (Participants) | 500
mg/kg | 3.49 [2.08 to 5.85]

9. Secondary Outcome: Impact of Remicade Location (Specialized Hospitals Versus Extramural Infusion Centers) on the Physical Component Summary Score (PCS)
Description: Participant's quality of life was measured by the short-form 36 (SF-36). The SF-36 is a survey with 36 questions. It is composed of the PCS & the Mental Component Summary Score (MCS). The SF-36 consisted of eight scaled scores, which were the weighted sums of the questions in their section. Each scale was directly transformed into a 0 (lowest level of functioning) - 100 (highest level of functioning) scale on the assumption that each question carried equal weight. The impact of the maintenance therapy location (specialized hospitals versus extramural infusion centers) was also examined.
Time Frame: 24 months maximum
Population: Remicade-naive participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 194 | 121
Score on a scale
  Baseline (n=194, n=121) | 31.25 (15.78) | 31.59 (16.81)
  Endpoint (after 9 infusions; n=125, n=13)) | 58.96 (22.26) | 42.46 (20.78)

10. Secondary Outcome: Impact of Remicade Location (Specialized Hospitals Versus Extramural Infusion Centers) on the MCS
Description: Participant's quality of life was measured by the short-form 36 (SF-36). The SF-36 is a survey with 36 questions. It is composed of the PCS & the MCS. The SF-36 consisted of eight scaled scores, which were the weighted sums of the questions in their section. Each scale was directly transformed into a 0 (lowest level of functioning) - 100 (highest level of functioning) scale on the assumption that each question carried equal weight. The impact of the maintenance therapy location (specialized hospitals versus extramural infusion centers) was also examined.
Time Frame: 24 months maximum
Population: Remicade-naive participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Remicade (Specialized Hospitals Only) | Remicade (Extramural Infusion Centers Only)
Number analyzed (Participants) | 194 | 124
Score on a scale
  Baseline (n=194, n=124) | 43.89 (17.98) | 45.12 (18.70)
  Endpoint (after 9 infusions; n=125, n=13) | 67.10 (20.96) | 46.18 (25.71)

ADVERSE EVENTS:
Arm/Group | Remicade (Specialized Hospitals & Extramural Infusion Centers)
Serious Adverse Events (participants affected / at risk) | 21/516
Other Adverse Events (participants affected / at risk) | 0/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remicade (Specialized Hospitals & Extramural Infusion Centers) (N=516)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Multi-organ failure (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (2)
Knee operation (Surgical and medical procedures) | 1 (1)
Wrist surgery (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No